CLINICAL TRIAL: NCT03206385
Title: Intensity Modulated Radiation Treatments Followed by A Stereotactic CyberKnife Boost Focused on the Gross Residual Pelvic Tumor Volume
Brief Title: IMRT Followed by CyberKnife Boost Focused on the Gross Residual Pelvic Tumor Volume
Acronym: Boost_Pelvis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Francois Baclesse, Luxembourg (Other)
Responsible Party: Sponsor
Other Study IDs: CK Boost Pelvis
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Pelvis Tumors
MeSH Terms: conditions — Pelvic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CK Boost pelvis
  Interventions: Radiation: Radiation treatment; Radiation: CK Boost Pelvis

INTERVENTIONS:
Radiation: Radiation treatment — 50 Gy will be delivered in the PTV 1 and 60 Gy in the PTV 2 simultaneously in 28 fractions (5 fractions a week) in no more than 40 days. Anytime, 95% of the prescribed dose will have to cover at least 90% of the PTV 1 and PTV 2.
Radiation: CK Boost Pelvis — Two high CyberKnife dose sessions will deliver a pelvic boost of 6.5 Gy each to the initial GTV or eventually to the residual GTV in case of too close vicinity of the OAR

SUMMARY:
The present register has been designed to confirm the hypothesis that while using high quality Intensity Modulated Radiation Techniques (IMRT) and a reduced external beam stereotactic boost component it would be possible to maintain the late severe toxicity rates under the 5 % level in situations where brachytherapy could not be proposed as a boost.

DETAILED DESCRIPTION:
This register concerned patients with any kind of non-resected pelvic cancer for which a brachytherapy Gross Tumor Volume (GTV) boost is non indicated.

1. Placement of fiducials First of all, fiducials will be placed near or inside the Gross Tumor Volume (GTV).
2. Radiation treatment The radiation treatment will be delivered by Varian Rapid ARC accelerators. 50 Gy will be delivered in the Planning Tumor Volume (PTV) 1 and 60 Gy in the PTV 2 simultaneously in 28 fractions (5 fractions a week) in no more than 40 days. Anytime, 95% of the prescribed dose will have to cover at least 90% of the PTV 1 and PTV 2.
3. CK Boost pelvis In the following 14 days after the external beam treatment, two high CyberKnife dose sessions will deliver a pelvic boost of 6.5 Gy each to the initial GTV or eventually to the residual GTV in case of too close vicinity of the organs at risk (OAR). This boost will be planned according to a recent paper, using a new CT scan and MRI scan for planimetric purposes. 95% of the prescribed dose will have to cover at least 90% of the PTV. The maximal CyberKnife tolerated doses to the OAR for a 6.5 Gy dose will be 5 Gy to 2cc of the bladder, rectum or sigmoid structures and 2.5 Gy to 5 cc of the small bowel. The protocol will not require a dose summation of the different steps of the treatment. The total duration of the whole treatment will have to be inferior to 55 days.

4 Follow-up The clinical follow up will be planed weekly during the radiation treatments, and at 2, 4 and 6 months thereafter. The patients will be then followed up every 4 months during the first 2 years and twice yearly thereafter.

A medical imaging using PET Scanner and MRI when possible will be performed at least at 6 months intervals during the first 2 years.

ELIGIBILITY:
Inclusion Criteria:

* any kind of locally advanced pelvic tumor, non-operable for any reason
* signed informed consent
* concomitant chemotherapy or hormonotherapy unless gemcitabine will not be contraindicated during the treatment

Exclusion Criteria:

* possibility to easily offer the patient a brachytherapy boost
* extra pelvic tumor dissemination above the L3 vertebra
* collagenoses
* any bowel tumor when the digestive tract is not definitely and locally bypassed
* any biologic targeted therapy or anti angiogenic therapy within the 6 weeks preceding the initiation of the radiation treatment, for the first 20 patients. This point will be revisited afterwards and will conduct to an amendment in case of protocol modification
* gemcitabine chemotherapy within the 6 weeks preceding the initiation of the radiation treatment or during the treatment
* hip prostheses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with any kind of non-resected pelvic cancer for which a brachytherapy Gross Tumor Volume (GTV) boost is non indicated
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-05-31 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Severe toxicity | follow up during 3 years after patient inclusion
  The objective is to confirm an expected toxicity level of severe toxicity < 5%

SECONDARY OUTCOMES:
Local clinical control rates | follow up during 3 years after patient inclusion
  Ths objective is to study the local control rates defined by a study panel board including at least a radiologist specially trained to review the imaging data after high radiation doses per fraction and the coordinator of the register, using PET Scanner, MRI and clinical data
Extra pelvic dissemination rates | follow up during 3 years after patient inclusion
  The objective is to study the dissemination data of the disease above the pelvis
Ability of the multi leaf collimator to better cover the PTVs and to help shortening the delivery times | follow up during 3 years after patient inclusion
  Using the different Conformal Index modalities, the objective is to compare the treatment planning with or without using the multi leaf collimator

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Francois Baclesse, Esch-sur-Alzette, SUD, Luxembourg

IPD SHARING:
Plan to Share IPD: No